CLINICAL TRIAL: NCT03621761
Title: A Randomized Controlled Trial of Telephone-delivered Cognitive Behavioral-therapy, Modafinil, and Combination Therapy of Both Interventions for Fatigue in Multiple Sclerosis
Brief Title: Cognitive Behavioral Therapy, Modafinil, or Both for Multiple Sclerosis Fatigue
Acronym: COMBO-MS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: University of Washington (Other); Patient-Centered Outcomes Research Institute (Other); National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Tiffany J. Braley, MD, MS, Assistant Professor of Neurology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00143319
Record Dates: First submitted 2018-08-03; First posted 2018-08-08 (Actual); Results first posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Multiple Sclerosis
Keywords: cognitive behavioral therapy; modafinil; Provigil; fatigue; MS
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Modafinil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Rater blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cognitive Behavioral Therapy (Active Comparator): 8 weekly telephone-based sessions and 2 booster sessions
  Interventions: Behavioral: Telephone-based Cognitive Behavioral Therapy
- Modafinil (Active Comparator): 50-400 mg per day (oral)
  Interventions: Drug: Modafinil
- Cognitive Behavioral Therapy + Modafinil (Active Comparator): Telephone-based cognitive behavioral therapy (8 weekly therapy sessions and 2 booster sessions) + Modafinil 50-400 mg per day (oral)
  Interventions: Behavioral: Telephone-based Cognitive Behavioral Therapy; Drug: Modafinil

INTERVENTIONS:
Behavioral: Telephone-based Cognitive Behavioral Therapy — Cognitive behavioral therapy (CBT) is a behavioral-based treatment that promotes effective self-management skills, including adaptive thought processes and behaviors (i.e. "coping skills"). CBT also commonly teaches goal-setting and behavioral activation strategies for engaging in physical, social, and other valued activities in the context of fatigue.
  Arms: Cognitive Behavioral Therapy; Cognitive Behavioral Therapy + Modafinil
Drug: Modafinil — Modafinil is a safe, well-tolerated and effective wake-promoting agent (oral medication) that is FDA-approved for the treatment of fatigue related to sleep disorders. Modafinil is also one of the most commonly used medications for multiple sclerosis related fatigue in clinical practice, with doses ranging from 50 - 400 mg per day, in divided doses (once to twice daily).
  Other Names: Provigil
  Arms: Cognitive Behavioral Therapy + Modafinil; Modafinil

SUMMARY:
This clinical trial will compare the effectiveness of 3 treatments for fatigue in Multiple Sclerosis: 1) a commonly used behavioral treatment strategy (telephone-based cognitive behavioral therapy), 2) a commonly used medication (modafinil), and 3) a combination of both therapies. Each participant will receive one of these 3 treatments for a total of 12 weeks. Hypotheses are that, at 12 weeks, treatment with combination therapy will overall lead to greater reductions in fatigue impact, fatigue severity, and fatigability compared to monotherapy, and that comorbid depression, sleep disturbances, and baseline disability level will be important effect modifiers that influence treatment effect and adherence.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinically definite Multiple Sclerosis (MS, all MS subtypes);
2. Age 18 years or older;
3. Presence of chronic, problematic fatigue that, in the opinion of the patient, has interfered with their daily activities for ≥ 3 months;
4. Average Fatigue Severity Scale (FSS) score greater or equal to 4 at screening.

Exclusion Criteria:

1. Current shift work sleep disorder, or narcolepsy diagnosed with polysomnography and multiple sleep latency test
2. History of MS relapse within the last 30 days prior to screening (participants will be considered eligible after the 30-day window);
3. Current stimulant or wake-promoting agent use (such as amantadine, modafinil, methylphenidate, or amphetamine) within 30 days of screening;
4. Pregnancy or breastfeeding;
5. Reliance on hormonal contraception AND concomitant unwillingness to use alternative non-hormonal means of birth control (spermicide or condoms) during the course of the study;
6. Current suicidal ideation (SI) with intent or plan;
7. Known hypersensitivity to modafinil or armodafinil or its inactive ingredients;
8. History of the following cardiovascular conditions: recent myocardial infarction (last 6 months prior to screening), unstable angina, left ventricular hypertrophy, mitral valve prolapse, NYHA class III or IV congestive heart failure;
9. History of prescription or illicit stimulant abuse (such as cocaine, amphetamine, methamphetamine);
10. Any other medical, neurological, or psychiatric condition that, in the opinion of the investigators, could affect participant safety or eligibility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany J Braley, MD, MS, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - The University of Michigan, Ann Arbor, Michigan
  - The University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krupp L. Fatigue is intrinsic to multiple sclerosis (MS) and is the most commonly reported symptom of the disease. Mult Scler. 2006 Aug;12(4):367-8. doi: 10.1191/135248506ms1373ed. No abstract available. PMID 16900749
- [Background] Lerdal A, Celius EG, Krupp L, Dahl AA. A prospective study of patterns of fatigue in multiple sclerosis. Eur J Neurol. 2007 Dec;14(12):1338-43. doi: 10.1111/j.1468-1331.2007.01974.x. Epub 2007 Sep 26. PMID 17903208
- [Background] Janardhan V, Bakshi R. Quality of life in patients with multiple sclerosis: the impact of fatigue and depression. J Neurol Sci. 2002 Dec 15;205(1):51-8. doi: 10.1016/s0022-510x(02)00312-x. PMID 12409184
- [Background] Krupp LB, Alvarez LA, LaRocca NG, Scheinberg LC. Fatigue in multiple sclerosis. Arch Neurol. 1988 Apr;45(4):435-7. doi: 10.1001/archneur.1988.00520280085020. PMID 3355400
- [Background] Smith MM, Arnett PA. Factors related to employment status changes in individuals with multiple sclerosis. Mult Scler. 2005 Oct;11(5):602-9. doi: 10.1191/1352458505ms1204oa. PMID 16193900
- [Background] Fisk JD, Pontefract A, Ritvo PG, Archibald CJ, Murray TJ. The impact of fatigue on patients with multiple sclerosis. Can J Neurol Sci. 1994 Feb;21(1):9-14. PMID 8180914
- [Background] Fisk JD, Ritvo PG, Ross L, Haase DA, Marrie TJ, Schlech WF. Measuring the functional impact of fatigue: initial validation of the fatigue impact scale. Clin Infect Dis. 1994 Jan;18 Suppl 1:S79-83. doi: 10.1093/clinids/18.supplement_1.s79. PMID 8148458
- [Background] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Background] Kroenke K, Spitzer RL, Williams JB. The Patient Health Questionnaire-2: validity of a two-item depression screener. Med Care. 2003 Nov;41(11):1284-92. doi: 10.1097/01.MLR.0000093487.78664.3C. PMID 14583691
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Derived] Braley TJ, Ehde DM, Alschuler KN, Little R, Ng YT, Zhai Y, von Geldern G, Chervin RD, Conroy D, Valentine TR, Romeo AR, LaRocca N, Hamade M, Jordan A, Singh M, Segal BM, Kratz AL. Comparative effectiveness of cognitive behavioural therapy, modafinil, and their combination for treating fatigue in multiple sclerosis (COMBO-MS): a randomised, statistician-blinded, parallel-arm trial. Lancet Neurol. 2024 Nov;23(11):1108-1118. doi: 10.1016/S1474-4422(24)00354-5. PMID 39424559

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician or clinic referral at two university medical centers, social media advertising, web site postings, email, letter, and phone calls to participants on our health registries. The first participant was enrolled on November 15, 2018 and the last participant was enrolled on June 2, 2021.
Pre-assignment Details: Of 343 enrolled participants, 336 met inclusion criteria and were randomized to treatment.
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy | Modafinil | Cognitive Behavioral Therapy + Modafinil
Started | 114 | 114 | 108
Week 8 Follow-up Timepoint | 111 | 111 | 105
Week 12 Follow-up Timepoint | 111 | 110 | 105
Week 24 Survey Timepoint | 111 | 110 | 105
Completed | 111 | 110 | 105
Not Completed | 3 | 4 | 3
Not completed — Lost to Follow-up | 1 | 1 | 2
Not completed — Withdrawal by Subject | 2 | 1 | 1
Not completed — Became Ineligible | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Therapy | Modafinil | Cognitive Behavioral Therapy + Modafinil | Total
Number analyzed (Participants) | 114 | 114 | 108 | 336
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (11.6) | 47.4 (11.7) | 49.1 (11.3) | 48.8 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 93 | 78 | 256
  Male | 29 | 21 | 30 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 6 | 4 | 8 | 18
  Ethnicity: Not Hispanic or Latino | 102 | 106 | 97 | 305
  Ethnicity: Unknown or Not Reported | 6 | 4 | 3 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 1 | 4
  Black or African American | 7 | 8 | 6 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  White | 96 | 98 | 92 | 286
  Other | 1 | 3 | 1 | 5
  Missing | 0 | 0 | 1 | 1
  Bi/Multi-Racial | 8 | 4 | 7 | 19
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 114 | 114 | 108 | 336
Modified Fatigue Impact Scale (MFIS) Score [Mean (Standard Deviation); unit: units on a scale] — The Modified Fatigue Impact Scale is a self-report survey that contains 21 items. Each item is rated 0-4. Higher scores indicate a greater impact of fatigue on a person's daily life. Total scores range from 0 - 84. Population: Baseline MFIS results (means/SD) are based on the number of participants who completed the entire survey at baseline. 10 participants in the CBT group, 8 participants in the combination group, and 7 in the modafinil group had incomplete survey results.
  units on a scale
    number analyzed (Participants) | 104 | 106 | 101 | 311
    (all) | 52.6 (13.7) | 53.2 (14.4) | 52.3 (14.1) | 52.7 (14.1)
Fatigue Intensity as Assessed by Self-reported Numerical Rating Scale (NRS) Score. [Mean (Standard Deviation); unit: units on a scale] — Fatigue intensity was assessed using a wearable monitor, the PRO-Diary (CamNtech) - a wrist-worn accelerometer-based activity monitor which also contains a self-report user interface.
  Using a 0-10 numerical rating scale, participants rated their fatigue intensity on the user-interface of the PRO-Diary four times each day, for 7 days, at baseline (pre-intervention). All scores over the 7 days are averaged to produce an aggregate fatigue intensity score. Higher scores indicate greater fatigue intensity. Population: 7 participants in the CBT group, 3 participants in the combination therapy group, and 3 participants in the modafinil group were missing baseline EMA fatigue intensity data.
  units on a scale
    number analyzed (Participants) | 107 | 111 | 105 | 323
    (all) | 9.2 (2.9) | 9.0 (3.2) | 8.8 (3.0) | 9.0 (3.0)
Fatigue Interference as Assessed by Self-reported Numerical Rating Scale (NRS) Score [Mean (Standard Deviation); unit: units on a scale] — Fatigue intereference was assessed using a wearable monitor, the PRO-Diary (CamNtech) - a wrist-worn accelerometer-based activity monitor which also contains a self-report user interface.
  Using a 0-10 numerical rating scale, participants rated their fatigue impact, and entered the score into the user-interface on the PRO-Diary four times each day, for 7 days, at baseline (pre-intervention). All scores over the 7 days are averaged to produce an aggregate fatigue interference score. Higher scores indicate greater fatigue interference. Population: 7 participants in the CBT group, 3 participants in the combination therapy group, and 3 participants in the modafinil group were missing baseline EMA fatigue interference data.
  units on a scale
    number analyzed (Participants) | 107 | 111 | 105 | 323
    (all) | 7.75 (3.15) | 7.33 (3.52) | 7.30 (3.32) | 7.5 (3.3)
Fatigability as Assessed by the Self-reported Fatigue Intensity Numerical Rating [Mean (Standard Deviation); unit: units on a scale] — Fatigability was assessed using a wearable monitor, the PRO-Diary (CamNtech) - a wrist-worn accelerometer-based activity monitor which also contains a self-report user interface. The fatigability score is calculated as the ratio of the self-reported fatigue intensity rating (using a 0-10 numerical rating score) divided by the participant's concurrent physical activity level (measured as the average number of activity counts per minute). All fatigability scores are averaged over the 7 days to create an aggregate fatigability score. Higher scores indicate greater fatigability. Population: 7 participants in the CBT group, 3 participants in the combination therapy group, and 3 participants in the modafinil group were missing baseline EMA fatigability data.
  units on a scale
    number analyzed (Participants) | 107 | 108 | 100 | 315
    (all) | 0.07 (0.04) | 0.07 (0.04) | 0.07 (0.07) | 0.07 (0.05)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Modified Fatigue Impact Scale (MFIS) Score
Description: The Modified Fatigue Impact Scale is a 21-item self-report survey. Each item is rated 0-4, Total scores range from 0-84. . Higher scores indicate a greater impact of fatigue on a person's activities. The primary outcome measure will be the mean within-subject difference between baseline and 12-week Modified Fatigue Impact Scale values (delta-MFIS), compared between the 3 treatment groups.
Time Frame: Baseline-12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy | Modafinil | Cognitive Behavioral Therapy + Modafinil
Number analyzed (Participants) | 114 | 114 | 108
score on a scale | -15.2 (11.9) | -16.0 (15.9) | -17.3 (16.2)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Cognitive Behavioral Therapy + Modafinil; Comparison of treatment effect of CBT monotherapy vs. combination therapy (reference) on total MFIS score, in linear regression models adjusted for age, sex, anxiety, pain, activity level, study site, and baseline MFIS score. Output reflects models that were imputed for missing data; Test type: Superiority; p = 0.3451, Regression, Linear; Slope = 1.7740
Statistical Analysis 2: Comparison: Modafinil vs Cognitive Behavioral Therapy + Modafinil; Comparison of treatment effect of modafinil monotherapy vs. combination therapy (reference) on total MFIS score, in linear regression models adjusted for age, sex, anxiety, pain, activity level, study site, and baseline MFIS score. Output reflects models that were imputed for missing data; Test type: Superiority; p = 0.4834, Regression, Linear; Slope = 1.3094

2. Secondary Outcome: Change in Fatigue Intensity as Assessed by Self-reported Numerical Rating Scale (NRS) Score.
Description: Fatigue intensity was assessed using a wearable monitor, the PRO-Diary (CamNtech) - a wrist-worn accelerometer-based activity monitor which also contains a self-report user interface. Using a 0-10 numerical rating scale, participants entered fatigue intensity ratings into the user-interface on the PRO-Diary 4 times each day, for 7 days, at baseline (pre-intervention) and at 12 weeks post-intervention. All scores over the 7 days were averaged to produce an aggregate fatigue intensity score. Higher scores indicate greater fatigue intensity. Change in fatigue intensity between baseline and 12 weeks was compared between the 3 treatment groups.
Time Frame: Baseline-12 weeks
Population: Some participants who completed the study did not complete their 12-week Pro-Diary entries.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy | Modafinil | Cognitive Behavioral Therapy + Modafinil
Number analyzed (Participants) | 88 | 91 | 93
units on a scale | -1.41 (2.43) | -1.69 (2.33) | -2.03 (2.82)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Cognitive Behavioral Therapy + Modafinil; Comparison of treatment effect of CBT monotherapy vs. combination therapy (reference) on change in EMA fatigue intensity NRS score, in complete case linear regression models adjusted for age, sex, anxiety, pain, activity level, study site, and baseline EMA fatigue intensity score; Test type: Superiority; p = 0.2570, Regression, Linear; Slope = 0.4077
Statistical Analysis 2: Comparison: Modafinil vs Cognitive Behavioral Therapy + Modafinil; Comparison of treatment effect of modafinil monotherapy vs. combination therapy (reference) on change in EMA fatigue intensity NRS score, in complete case linear regression models adjusted for age, sex, anxiety, pain, activity level, study site, and baseline EMA fatigue intensity score; Test type: Superiority; p = 0.5017, Regression, Linear; Slope = -0.2452

3. Secondary Outcome: Change in Fatigue Interference as Assessed by Self-reported Numerical Rating Scale (NRS) Score
Description: Fatigue interference will be assessed using a wearable monitor, the PRO-Diary (CamNtech) - a wrist-worn accelerometer-based activity monitor which also contains a self-report user interface. Using a 0-10 numerical rating scale, participants entered fatigue interference ratings into the user-interface on the PRO-Diary 4 times each day, for 7 days, at baseline (pre-intervention) and at 12 weeks post-intervention. All scores over the 7 days were averaged to produce an aggregate fatigue impact score. Higher scores indicate greater fatigue impact. Change in fatigue interference between baseline and 12 weeks will be compared between the 3 treatment groups.
Time Frame: Baseline-12 weeks
Population: A few participants in each arm who stayed in the study, did not complete the NRS Survey at 12 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy | Modafinil | Cognitive Behavioral Therapy + Modafinil
Number analyzed (Participants) | 88 | 91 | 93
score on a scale | -1.41 (2.60) | -1.73 (2.52) | -1.78 (2.98)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Cognitive Behavioral Therapy + Modafinil; Comparison of treatment effect of CBT monotherapy vs. combination therapy (reference) on change in EMA fatigue interference NRS score, in complete case linear regression models adjusted for age, sex, anxiety, pain, activity level, study site, and baseline EMA fatigue interference score; Test type: Superiority; p = 0.154, Regression, Linear; Slope = 0.095
Statistical Analysis 2: Comparison: Modafinil vs Cognitive Behavioral Therapy + Modafinil; Comparison of treatment effect of modafinil monotherapy vs. combination therapy (reference) on change in EMA fatigue interference NRS score, in complete case linear regression models adjusted for age, sex, anxiety, pain, activity level, study site, and baseline EMA fatigue interference score; Test type: Superiority; p = 0.610, Regression, Linear; Slope = 0.034

4. Secondary Outcome: Change in Fatigability as Assessed by the Self-reported Fatigue Intensity Numerical Rating Scale (NRS) Score and Physical Activity Level
Description: Fatigability will be assessed using a wearable monitor, the PRO-Diary (CamNtech) - a wrist-worn accelerometer-based activity monitor which also contains a self-report user interface. The fatigability score will be calculated as the ratio of the self-reported fatigue intensity rating (using a 0-10 numerical rating score) divided by the participant's concurrent physical activity level (measured as the average number of activity counts per minute via actigraphy). All fatigability scores will be averaged over the 7 days to create an aggregate fatigability score. Higher scores indicate greater fatigability. Change in fatigability between baseline and 12 weeks will be compared between the 3 treatment groups.
Time Frame: Baseline-12 weeks
Population: Some participants in the study did not complete their 12-week Pro-Diary entries.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Cognitive Behavioral Therapy | Modafinil | Cognitive Behavioral Therapy + Modafinil
Number analyzed (Participants) | 83 | 83 | 86
score | -0.0041 (0.0476) | -0.0175 (0.0320) | -0.0075 (0.0404)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Cognitive Behavioral Therapy + Modafinil; Comparison of treatment effect of CBT monotherapy vs. combination therapy (reference) on change in fatigability score, in complete case linear regression models adjusted for age, sex, anxiety, pain, activity level, study site, and baseline fatigability score; Test type: Superiority; p = 0.4955, Regression, Linear; Slope = 0.00427
Statistical Analysis 2: Comparison: Modafinil vs Cognitive Behavioral Therapy + Modafinil; Comparison of treatment effect of modafinil monotherapy vs. combination therapy (reference) on change in fatigability score, in complete case linear regression models adjusted for age, sex, anxiety, pain, activity level, study site, and baseline fatigability score; Test type: Superiority; p = 0.1333, Regression, Linear; Slope = -0.00948

ADVERSE EVENTS:
Time Frame: 25 weeks, AE data was collected for 25 weeks from consent, in line with 24 week exploratory outcome measures.
Arm/Group | Cognitive Behavioral Therapy | Modafinil | Cognitive Behavioral Therapy + Modafinil
All-Cause Mortality (participants affected / at risk) | 0/114 | 1/114 | 0/108
Serious Adverse Events (participants affected / at risk) | 1/114 | 4/114 | 1/108
Other Adverse Events (participants affected / at risk) | 1/114 | 12/114 | 19/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cognitive Behavioral Therapy (N=114) | Modafinil (N=114) | Cognitive Behavioral Therapy + Modafinil (N=108)
MS relapse/exacerbation (Nervous system disorders) | 1 | 2 | 1
Benign paroxysmal vertigo (Nervous system disorders) | 1 | 0 | 0
Cerebrospinal fluid leakage (Blood and lymphatic system disorders) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Localized edema (Immune system disorders) | 0 | 0 | 1
Pneumonia (Nervous system disorders) | 0 | 0 | 1
Trigeminal neuralgia pain (Nervous system disorders) | 0 | 0 | 1
Surgical/Medical procedure (Surgical and medical procedures) | 1 | 4 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cognitive Behavioral Therapy (N=114) | Modafinil (N=114) | Cognitive Behavioral Therapy + Modafinil (N=108)
Insomnia (Nervous system disorders) | 0 | 8 | 8
Anxiety (Nervous system disorders) | 0 | 3 | 9
Headache (Nervous system disorders) | 1 | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT03621761/Prot_SAP_001.pdf